CLINICAL TRIAL: NCT04929106
Title: Physical Activity With Tailored mHealth Support for Individuals With Intellectual Disability - a Mixed Method Pilot Study
Brief Title: Physical Activity, mHealth and Intellectual Disability - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/1770
Record Dates: First submitted 2021-06-07; First posted 2021-06-18 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2021-06

CONDITIONS: Intellectual Disability
Keywords: Intellectual Disability; Physical Activity; Technology; mHealth
MeSH Terms: conditions — Intellectual Disability; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHealth intervention (Experimental): Tailored physical activity program with motivational mobile health support on everyday levels of physical activity
  Interventions: Device: mHealth support tool

INTERVENTIONS:
Device: mHealth support tool — The final app is named Active Leisure and consists of an advanced activity planner based on the platform developed by the ideal company Smart Cognition AS. The app offers different interface options (symbols only, easy to read text, plain text, and read aloud). The activity planner will mostly be used by the individual with IDs and a support person (caregiver or health care provider). After completing an activity, a simple reward is available (e.g., a smiling face or to share a picture with other users of the app). The use of tailored communication through personalization: the use of individuals first name in the activity planner, adaptation: individually chosen activities, adjusted communication (symbols, easy-to-read text or plain text), preparation and planning, and feedback: rewarding and positive feedback (after activities have been performed) is expected to increase motivation, and thereby lead to higher levels of PA.

SUMMARY:
The main objective of this pilot study is to assess distant procedures, study experiences and feasibility of a planned randomized controlled trial investigating the use of a mHealth support tool on physical activity for individuals with intellectual disability.

DETAILED DESCRIPTION:
For individuals with intellectual disability (ID) with low physical activity (PA) levels, new methods to increase participation in physical activity are needed. Motivation for participation in PA should include both individuals with ID, family members and staff, and it should work in a supportive way to strengthen mastery experiences. Technology-based interventions have not yet been explored extensively.

The study objective is to assess feasibility of procedures for a distant, COVID-19-secure intervention, study pre-treatment expectations and experiences of participants and their caregivers. In addition, the study will explore the effectiveness of an individually tailored PA program with motivational mobile health support on everyday levels of PA, goal setting and self-efficacy in a PA setting for youth and adults with intellectual disabilities.

The current protocol concerns the conducting of a mixed method pilot study to test intervention procedures of a planned complex randomised controlled trial, with steps per day as main outcome. Ten participants with intellectual disability are included. Assessment are at baseline, follow-up after 4 weeks and 12 weeks. Goal attainment scale will be used together with the introduction of an activity planner application named Active Leisure as the intervention. Feasibility and acceptance of procedures, activity measures and questionnaires are assessed.

The present trial will investigate how modern technology and e-health can be used in the promotion of PA in individuals with IDs. The study has potentially important implications for both individuals with IDs and their support networks. If successful, the project will provide a simple and accessible solution for promoting PA in individuals with IDs.

ELIGIBILITY:
Inclusion Criteria:

* Low physical activity levels: determined with the question "How much of your leisure time have you been physically active in the last year?"
* Diagnosis of intellectual disability (mild, moderate, severe, or profound)
* Aged 16-60 years old
* Ability to participate in the intervention
* Ability to walk with or without support
* Able to provide written informed consent or written informed consent can be obtained from a representative

Exclusion Criteria:

* Medical contraindications for participation in programs with increased exercise, as advised by the primary care or ID specialist physician
* High level of physical activity
* Inability to provide written informed consent and written informed consent cannot be obtained from a representative

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in steps per day | Baseline, 4 weeks, 12 weeks
  Objectively measured physical activity assessed by steps per day measured with a wrist-worn commercial accelerometer (Fitbit Versa, Fitbit, Inc., San Francisco, CA, USA). The device will assess level of physical activity and sedentary time. The watch will show a neutral screen during baseline and follow-up assessments. Level of physical activity will be measured for 7 days at each assessment, with a minimum of 3 consecutive days of measurement because previous research has shown that 3 days of physical activity can predict weekly level of physical activity.

SECONDARY OUTCOMES:
Minutes of moderate physical acitivty | Baseline, 4 weeks, 12 weeks
  Secondary PA outcomes are minutes of moderate PA per day measured with a wrist-worn commercial fitness tracker (Fitbit Versa, Fitbit, Inc., San Francisco, CA, USA).
Physical activity levels | Baseline, 4 weeks, 12 weeks
  The International Physical Activity Questionnaire - Short Form, adapted to measure physical activity using proxy respondents will be used. The International Physical Activity Questionnaire - Short Form is a 7-item questionnaire that assesses PA in the past 7 days at 4 intensity levels: 1) vigorous-intensity activity, such as aerobics, 2) moderate-intensity activity, such as leisure cycling, 3) walking, and 4) sitting.
Behavioral problems | Baseline, 4 weeks, 12 weeks
  The Aberrant Behavior Checklist-Community (ABC-C) is a questionnaire designed to assess challenging behavior in children, youth, and adults with IDs. The checklist consist of 58 items divided into 5 subscales: irritability, lethargy, stereotypy, hyperactivity, and inappropriate speech. It is a proxy measure requiring knowledge of the person with ID. Each item is scored on a scale of 0-3 (3 indicating the most severity). The questionnaire has been validated for use in a Norwegian population with neurodevelopmental disabilities.
Social support for physical activity and self-efficacy in a physical activity setting | Baseline, 4 weeks, 12 weeks
  The Self-Efficacy/Social Support for Activity for persons with Intellectual Disability scale (SE/SS-AID) is a questionnaire consisting of four subscales. One subscale measures self-efficacy for overcoming barriers to leisure physical activity. The last three subscales measure social support for leisure activity from family members, care staff, and friends for individuals with intellectual disabilities. The scale has been validated for self-reporting from individuals with mild to moderate intellectual disability and for use by proxy respondents. The questionnaire will be translated into the Norwegian language using standard guidelines.
Satisfaction with life | Baseline, 4 weeks, 12 weeks
  This study will use the satisfaction with life scale developed by Bergström & Hochwälder, which was designed to assess satisfaction with the home environment and leisure time in individuals with mild to moderate intellectual disability. The scale has four factors: 1) satisfaction with housing environment, 2) satisfaction with life, 3) satisfaction with meals, and 4) satisfaction with recreational activities. Items are read aloud by a researcher and answered by participants with three response options: "good" (happy face = 2), "in between" (neutral face = 1), or "bad" (sad face = 0). In the current study, the scale is used to control for adverse effects.
Goal Attainment | Introduced together with intervention, 1 week after baseline
  Goal attainment scaling will be used to identify self-management goals that participants would like to achieve. The questionnaire will be filled out by the researcher, with participants and proxy respondents present. Goal attainment scaling involves several steps. Goals are selected by each individual, and observable behavior that reflects a degree of goal attainment is defined. The participant's pre-treatment or baseline levels are defined in terms of the goal. Five different goal attainment levels are used, ranging from "no change" to "much better than expected outcome" (numbered -2 to +2). Follow-up times for participant evaluation are set (presumably after 3 and 6 months). Goal attainment is evaluated after the defined time interval. At the end, the overall attainment score for all goals are calculated. In this study we will define up to three goals for PA.

CONTACTS AND LOCATIONS:
Overall Officials: Audny Anke, Prof. MD, Study Director — University Hospital of North Norway, UiT Artic University of Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michalsen H, Wangberg SC, Hartvigsen G, Jaccheri L, Muzny M, Henriksen A, Olsen MI, Thrane G, Jahnsen RB, Pettersen G, Arntzen C, Anke A. Physical Activity With Tailored mHealth Support for Individuals With Intellectual Disabilities: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jun 29;9(6):e19213. doi: 10.2196/19213. PMID 32437328
- [Result] Michalsen H, Wangberg SC, Anke A, Hartvigsen G, Jaccheri L, Arntzen C. Family members and health care workers' perspectives on motivational factors of participation in physical activity for people with intellectual disability: A qualitative study. J Intellect Disabil Res. 2020 Apr;64(4):259-270. doi: 10.1111/jir.12716. Epub 2020 Jan 24. PMID 31981261
- [Derived] Michalsen H, Wangberg SC, Hartvigsen G, Henriksen A, Pettersen G, Jaccheri L, Jahnsen RB, Thrane G, Arntzen C, Anke A. mHealth Support to Stimulate Physical Activity in Individuals With Intellectual Disability: Protocol for a Mixed Methods Pilot Study. JMIR Res Protoc. 2022 Sep 15;11(9):e37849. doi: 10.2196/37849. PMID 36107473